CLINICAL TRIAL: NCT04129125
Title: A Prospective, Multi-center, Open Label and Single Arm Clinical Investigation to Evaluate the Safety and Efficacy of Using the Zoom Reperfusion System in Thrombectomy Procedures to Treat Acute Ischemic Stroke Patients
Brief Title: The Imperative Trial: Treatment of Acute Ischemic Stroke With the Zoom Reperfusion System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperative Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICI-001
Record Dates: First submitted 2019-09-27; First posted 2019-10-16 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke; Acute Stroke
Keywords: stroke, thrombectomy, Zoom, aspiration, reperfusion, mRS
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, open-label with independent outcome assessments.
Masking Description: Reperfusion will be graded by an independent core lab that is not an enrolling investigational site.
  Neurological Outcome Assessors (NIHSS assessment): Neurological outcome assessors who will perform post-procedure 24-hour NIHSS assessments are NIHSS certified team members not performing the thrombectomy procedure and with no financial conflict of interest with Imperative Care, Inc.
  Functional Outcome Assessors (mRS assessment): Functional outcome assessors who will perform post-procedure assessments are part of achieving unbiased study objectives. They will not have access to patient data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Zoom Reperfusion System (Experimental): The subject will undergo the endovascular thrombectomy procedure under general anesthesia or conscious sedation. The Imperative Care .088" Catheter will be used to gain access to the vasculature and direct aspiration of the clot will be attempted where feasible. The Zoom Reperfusion System must be the initial and primary device used to remove thrombus.
  Interventions: Device: Zoom Reperfusion System

INTERVENTIONS:
Device: Zoom Reperfusion System — Thrombectomy

SUMMARY:
The trial is designed to assess the safety and efficacy of using the Zoom Reperfusion System in subjects diagnosed with acute ischemic stroke and undergoing a thrombectomy procedure within 8 hours of last known well.

DETAILED DESCRIPTION:
Each year 17 million people suffer stroke worldwide. According to the World Stroke Organization, stroke has become the second cause of death and disability worldwide. In the United States, every year, more than 795,000 people have a stroke. Given the large-scale challenges of curing stroke, prevention and treatments for stroke are much needed. Ischemic stroke is treatable in many patients if they have early access to viable treatments.

This trial is a prospective, multicenter, open-label, single-arm trial designed to assess the potential treatment benefits of using the Imperative Care 0.088" Catheters in conjunction with the other devices in the Zoom Reperfusion System to restore blood flow in patients with acute ischemic stroke secondary to intracranial large vessel occlusive disease. The Zoom Reperfusion System includes the Imperative Care 0.088" Catheters, the Zoom Reperfusion Catheters (0.035" to 0.071" Catheters), Zoom Aspiration Tubing, and Zoom Aspiration Pump. The trial will assess reperfusion success using the mTICI scores in the absence of any rescue therapy, reperfusion time, first-pass success, and functional independence including a quality-of-life assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. NIHSS >=6
3. The operator feels that the stroke can be treated with endovascular thrombectomy approaches and the interventionalist estimates that groin puncture can be achieved within 8 hours from time last seen well
4. Pre-event mRS scale 0-1
5. Large vessel occlusion of the intracranial internal carotid artery (ICA), middle cerebral artery (MCA)-M1 or M2 segments, basilar, or vertebral arteries as evidenced by MRA or CTA
6. For strokes in anterior circulation, ASPECTS >=6; For strokes in posterior circulation, pc-ASPECTS >=8
7. Non-contrast CT/CTA or MRI/MRA for trial eligibility performed or repeated at treating stroke center or outside medical facility within 2 hours of treatment initiation
8. If indicated per American Heart Association clinical guidelines, thrombolytic therapy should be administered as soon as possible
9. Consenting requirements met according to local IRB or Ethics Committee

Exclusion Criteria:

1. Female known to be pregnant at time of admission
2. Patient has suffered a stroke in the past 3 months
3. Presence of an existing or pre-existing large territory infarction
4. Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluation, e.g., dementia with prescribed anti-cholinesterase inhibitor
5. Known history of severe contrast allergy or absolute contraindication to iodinated contrast
6. Clinical history, past imaging or clinical judgement suggest that the intracranial occlusion is chronic
7. Life expectancy of less than 6 months prior to stroke onset
8. Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories
9. Subject participating in another clinical trial involving an investigational device or drug
10. Known cancer with metastases
11. Evidence of active systemic infection
12. Any known hemorrhagic or coagulation deficiency

    Imaging Exclusion Criteria:
13. Evidence of intracranial hemorrhage on CT/MRI
14. CTA or MRA evidence of carotid stenosis requiring treatment for intracranial access
15. Excessive vascular access tortuosity or target vessel size that will likely prevent endovascular access with the Imperative Care 0.088" ID Catheters
16. Intracranial stent implanted in the same vascular territory that would preclude the safe deployment/removal of the thrombectomy devices
17. Occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior circulation/vertebrobasilar system) as confirmed on CTA/MRA, or clinical evidence of bilateral strokes or strokes in multiple territories as determined by the treating physician
18. Significant mass effect with midline shift as confirmed on CT/MRI
19. Evidence of intracranial tumor (except small meningioma defined as ≤ 3cm and asymptomatic) as confirmed on CT/MRI
20. Angiographic evidence of pre-existing arterial injury, e.g., carotid dissection, complete cervical carotid occlusion, or vasculitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raul G Nogueira, MD, Principal Investigator — University of Pittsburgh; Reade A De Leacy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; William J Mack, MD, Principal Investigator — University of Southern California; Emir Deljkich, Study Director — Imperative Care, Inc.
Locations (28):
- United States (28):
  - Radiology of Huntsville, Huntsville, Alabama
  - Carondelet Neurological Institute St. Joseph's Hospital, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - John Muir Health, Walnut Creek, California
  - Baptist Health, Jacksonville, Florida
  - University of Miami / Jackson Memorial Hospital, Miami, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Tampa General Hospital / University of South Florida, Tampa, Florida
  - Grady Memorial Hospital / Emory University, Atlanta, Georgia
  - Ochsner Health, New Orleans, Louisiana
  - Spectrum Health, Grand Rapids, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Cooper University Health Care, Camden, New Jersey
  - The State University of New York at Buffalo, Buffalo, New York
  - Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oklahoma University, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - University of Pennsylvania, Pittsburgh, Pennsylvania
  - Prisma Health - Upstate, Greenville, South Carolina
  - Erlanger Health System: Tennessee Interventional and Imaging Associates, Chattanooga, Tennessee
  - Semmes Murphey Foundation / Methodist University Hospital, Memphis, Tennessee
  - Baylor Scott and White Research Institute, Dallas, Texas
  - Valley Baptist Medical Center, Harlingen, Texas
  - The University of Texas Health Science Center at Houston // Memorial Hermann Health System, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mack W, De Leacy RA, Grossberg JA, Majidi S, Tomalty RD, Mokin M, Vargas J, Cucchiara BL, Snyder KV, Mascitelli J, Parada V, Shakir HJ, Rosenbaum-Halevi D, Aghaebrahim A, Hoit D, Yim B, Tenser MS, Al-Bayati AR, Milburn JM, Nimjee SM, Haranhalli N, Nahhas M, Shaff D, Layton KF, Beaty N, Starke RM, Hawk H, Haussen DC, Pabaney A, Kellner CP, Nogueira RG. Stroke thrombectomy with a novel reperfusion system including a 0.088'' aspiration catheter: the Imperative Trial. J Neurointerv Surg. 2025 Jul 22:jnis-2025-023719. doi: 10.1136/jnis-2025-023719. Online ahead of print. PMID 40695608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2021 and March 2024, participants were recruited across 26 institutions in the United States.
Groups:
- Zoom Reperfusion System: Aspiration thrombectomy using Zoom Reperfusion System
Period: Overall Study
Arm/Group | Zoom Reperfusion System
Started | 328 (A total of 328 participants provided informed consent and were considered enrolled in the study. Of these, 263 subjects were site-assessed as meeting study inclusion and exclusion criteria (ITT population). There were only three (3) cases where treatment with the study device was not attempted as the first therapeutic approach and these cases were excluded from the ITT population, resulting in a mITT population consisting of 260 subjects.)
Completed | 260 (modified intent-to-treat population)
Not Completed | 68
Not completed — Participants did not meet eligibility criteria | 65
Not completed — Study device was not used | 3

BASELINE CHARACTERISTICS:
Population: modified intent-to-treat population
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 106
  >=65 years | 154
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [59 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 211
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  United States | 260

OUTCOME MEASURES:

1. Primary Outcome: ITT Cohort: Rate of Core Lab-adjudicated Reperfusion Success
Description: Reperfusion success was defined as achieving a modified Treatment in Cerebral Infarction (mTICI) score of ≥2b within three or fewer passes using the study device and without rescue therapy (e.g., additional thrombectomy devices or intra-arterial lytics). The mTICI scale ranges from 0 to 3, with higher scores indicating better reperfusion: 0 = no perfusion, 1 = minimal perfusion, 2a = partial (<50%), 2b = substantial (≥50%), 2c = near complete, 3 = complete. This measure reports the number of participants who achieved mTICI ≥2b under these criteria as adjudicated by an independent core lab.
Time Frame: Intraprocedural
Population: ITT Cohort: Post thrombectomy imaging available for core lab adjudication.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 259
Participants | 216
Statistical Analysis 1: Comparison: Zoom Reperfusion System; The FDA agreed performance goal for the primary efficacy endpoint was for the lower bound of the two-sided 95% CI to be >69%; Test type: Other — The study sample size of 260 subjects was selected to have at least 90 percent power for primary safety and efficacy endpoints and all-cause mortality; p < 0.0001, Fisher Exact — The p-value a priori threshold for statistical significance was <0.025; Event rate = 83.4, 95% CI 2-sided [78 to 88]

2. Primary Outcome: ITT Cohort: Rate of Symptomatic Intracranial Hemorrhage (sICH), as Independently Adjudicated by Core Lab and Safety Board
Description: Rate of symptomatic intracranial hemorrhage (sICH), as independently adjudicated by the core lab and the independent safety board
Time Frame: 24-hour post-procedure
Population: ITT Cohort: Post-thrombectomy imaging available for core lab and independent safety board adjudication
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 260
Participants | 5
Statistical Analysis 1: Comparison: Zoom Reperfusion System; The FDA agreed performance goal for the primary safety endpoint was for the observed rate to be ≤6.0%; Test type: Other — [test comment as in outcome 1, analysis 1]; Event rate = 1.9, 95% CI 2-sided [0.6 to 4.4]

3. Primary Outcome: FDA Clearance Cohort: Rate of Core Lab-adjudicated Reperfusion Success
Description: as for outcome 1
Time Frame: Intraprocedural
Population: The FDA Clearance Cohort comprises participants in whom concomitant dual aspiration was used (e.g., 0.088" ID and a smaller ID catheter)
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 211
Participants | 177
Statistical Analysis 1: Comparison: Zoom Reperfusion System; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0001, Fisher Exact — The p-value a priori threshold for statistical significance was <0.025; Event rate = 84, 95% CI 2-sided [78 to 89]

4. Primary Outcome: FDA Clearance Cohort: Rate of Symptomatic Intracranial Hemorrhage (sICH), as Independently Adjudicated by Core Lab and Safety Board
Description: as for outcome 2
Time Frame: 24-hour post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 211
Participants | 2
Statistical Analysis 1: Comparison: Zoom Reperfusion System; The FDA agreed performance goal for the primary safety endpoint was for the observed rate to be ≤6.0%; Test type: Other — [test comment as in outcome 1, analysis 1]; Event rate = 0.9, 95% CI 2-sided [0.1 to 3.4]

5. Primary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of Core Lab-adjudicated Reperfusion Success
Description: as for outcome 1
Time Frame: Intraprocedural
Population: FDA Clearance Cohort - Covariate Analysis for Distal ICA/M1 Occlusions. Procedural imaging was not available for one (1) participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 145
Participants | 125

6. Primary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of Symptomatic Intracranial Hemorrhage (sICH), as Independently Adjudicated by Core Lab and Safety Board
Description: as for outcome 2
Time Frame: 24-hour post-procedure
Population: FDA Clearance Cohort - Covariate Analysis for Distal ICA/M1 Occlusions; Based on available imaging and NIHSS.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 146
Participants | 1

7. Secondary Outcome: ITT Cohort: Time to Achieve mTICI Score ≥ 2b
Description: The time from groin puncture to mTICI (modified treatment in cerebral infarction) score ≥ 2b
  mTICI range: 0 to 3; higher score means better reperfusion
Time Frame: Intraprocedural
Population: ITT Cohort
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 260
minutes | 19 [13 to 30]

8. Secondary Outcome: ITT Cohort: Rate of mTICI Score 3 Reperfusion
Description: Independent core lab-adjudicated reperfusion success, defined as modified treatment in cerebral infarction (mTICI) score = 3 within three or fewer passes with the study device, without using rescue therapy (e.g., additional thrombectomy devices or intra-arterial lytics)
  mTICI range: 0 to 3; higher score means better reperfusion
Time Frame: Intraprocedural
Population: ITT Cohort: Post thrombectomy imaging available for core lab adjudication
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 259
Participants | 78

9. Secondary Outcome: ITT Cohort: Rate of First Pass Success
Description: Independent core lab-adjudicated modified treatment in cerebral infarction (mTICI) score ≥2b after the first pass with the study device
  mTICI range: 0 to 3; higher score means better outcome
Time Frame: Intraprocedural
Population: ITT Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 259
Participants | 148

10. Secondary Outcome: ITT Cohort: Rate of mTICI Score 2c Reperfusion
Description: Independent core lab-adjudicated reperfusion success, defined as modified treatment in cerebral infarction (mTICI) score ≥2c within three or fewer passes with the study device, without using rescue therapy (e.g., additional thrombectomy devices or intra-arterial lytics)
  mTICI range: 0 to 3; higher score means better outcome
Time Frame: Intraprocedural
Population: ITT Cohort: Post thrombectomy imaging available for core lab adjudication.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 259
Participants | 147

11. Secondary Outcome: ITT Cohort: Rate of Functional Independence
Description: The proportion of patients achieving modified Rankin Scale (mRS) score ≤2 using the primary treatment modality, evaluated by certified assessors
  The mRS scale ranges from 0 (no symptoms) to 5 (severe disability), with an additional category of 6 for death
Time Frame: 90-days post-procedure
Population: ITT Cohort: Subjects with completed mRS assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 244
Participants | 133

12. Secondary Outcome: ITT Cohort: Quality of Life Assessment
Description: The Stroke Impact Scale (SIS) is a self-reported questionnaire assessing quality of life in 8 domains: Strength, Memory and Thinking, Emotion, Communication, ADL/IADL, Mobility, Hand Function, and Participation/Role Function. Each domain is scored from 0 to 100, with higher scores indicating better function and less impact of stroke. Scores are calculated by averaging item responses in each domain and transforming to a 0-100 scale. A separate recovery score from 0 (no recovery) to 100 (full recovery) reflects the patient's overall perception of recovery. Domain scores are not combined into a total score.
Time Frame: 90 days post-procedure
Population: ITT Cohort: Participants that completed the SIS Questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 185
score on a scale
  Overall Recovery | 71.5 (25.8)
  Strength | 71 (27.9)
  Memory and Thinking | 79.9 (21.9)
  Emotion | 78.9 (17.9)
  Communication | 85 (22.6)
  Activities of Daily Living or Instrumental Activities of Daily Living | 76.3 (28.5)
  Mobility | 71.5 (29.5)
  Hand Function | 68.9 (36)
  Participation/Role Function | 70.1 (29.7)

13. Secondary Outcome: ITT Cohort: Rate of All-Cause Mortality
Description: Rate of 90-day all-cause mortality
Time Frame: 90 days post-procedure
Population: ITT Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 260
Participants | 33
Statistical Analysis 1: Comparison: Zoom Reperfusion System; The FDA agreed performance goal for the all-cause mortality endpoint was for the observed rate to be ≤20.3%; Test type: Other — [test comment as in outcome 1, analysis 1]; Event rate = 12.7, 95% CI 2-sided [8.5 to 16.7] — Event and CI estimated using Kaplan-Meier method

14. Secondary Outcome: ITT Cohort: Rate of All Intracranial Hemorrhage (ICH)
Description: Independent core lab adjudicated rate of all ICH at 24-hour post-procedure
Time Frame: 24-hour post-procedure
Population: ITT Cohort: Post thrombectomy imaging available for core lab adjudication.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 259
Participants | 53

15. Secondary Outcome: ITT Cohort: Rate of Embolization in New Territory (ENT)
Description: Rate of participants with embolism into a new territory (ENT) as evidenced by new occlusions noted post-procedure or new infarcts identified on 24-hour imaging that are remote to the vascular territory impacted by the index stroke
Time Frame: 24-hour post-procedure
Population: ITT Cohort: Subjects with completed ENT assessment forms
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 246
Participants | 2

16. Secondary Outcome: ITT Cohort: Rate of Serious Adverse Device Effects (SADEs)
Description: Independent Safety Board adjudicated device-related serious adverse device events within 90 days post-procedure
Time Frame: 90 days post-procedure
Population: ITT Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 260
Participants | 5

17. Secondary Outcome: ITT Cohort: Rate of Serious Adverse Events
Description: All serious adverse events through 90 days post-procedure.
Time Frame: 90 days post-procedure
Population: ITT Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 260
Participants | 95

18. Secondary Outcome: FDA Clearance Cohort: Time to Achieve mTICI Score ≥ 2b
Description: as for outcome 7
Time Frame: Intraprocedural
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 211
minutes | 19 [12 to 29]

19. Secondary Outcome: FDA Clearance Cohort: Rate of mTICI Score 3 Reperfusion
Description: Independent core lab-adjudicated reperfusion success, defined as modified treatment in cerebral infarction (mTICI) score = 3 within three or fewer passes with the study device, without using rescue therapy (e.g., additional thrombectomy devices or intra-arterial lytics)
  mTICI range: 0 to 3; higher score means better outcome
Time Frame: Intraprocedural
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Zoom Reperfusion System: Thrombectomy using Zoom Reperfusion System
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 211
Participants | 65

20. Secondary Outcome: FDA Clearance Cohort: Rate of First Pass Success
Description: as for outcome 9
Time Frame: Intraprocedural
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 211
Participants | 128

21. Secondary Outcome: FDA Clearance Cohort: Rate of mTICI Score 2c Reperfusion
Description: Independent core lab-adjudicated reperfusion success, defined as modified treatment in cerebral infarction (mTICI) score ≥2c within three or fewer passes with the study device, without using rescue therapy (e.g., additional thrombectomy devices or intra-arterial lytics)
  mTICI range: 0 to 3; higher score means better reperfusion
Time Frame: Intraprocedural
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 211
Participants | 124

22. Secondary Outcome: FDA Clearance Cohort: Rate of Functional Independence
Description: as for outcome 11
Time Frame: 90-days post-procedure
Population: Subjects with completed mRS assessments. The FDA Clearance Cohort comprises participants in whom concomitant dual aspiration was used (e.g., 0.088" ID and a smaller ID catheter).
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 198
Participants | 110

23. Secondary Outcome: FDA Clearance Cohort: Quality of Life Assessment
Description: as for outcome 12
Time Frame: 90-days post-procedure
Population: The FDA Clearance Cohort comprises participants in whom concomitant dual aspiration was used (e.g., 0.088" ID and a smaller ID catheter). The sample size includes participants who completed Stroke Impact Scale (SIS) Questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 146
score on a scale
  Overall Recovery | 72.7 (25.7)
  Strength | 72.4 (27.3)
  Memory and Thinking | 79.8 (22.6)
  Emotion | 79.2 (18)
  Communication | 85.7 (21.7)
  Activities of Daily Living or Instrumental Activities of Daily Living | 77.8 (28.3)
  Mobility | 73.8 (28.4)
  Hand Function | 70.5 (34.9)
  Participation/Role Function | 70.8 (29.9)

24. Secondary Outcome: FDA Clearance Cohort: Rate of All-Cause Mortality
Description: Rate of 90-day all-cause mortality
Time Frame: 90-days post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 211
Participants | 26
Statistical Analysis 1: Comparison: Zoom Reperfusion System; The FDA agreed performance goal for the primary safety endpoint was for the observed rate to be ≤20.3%; Test type: Other — [test comment as in outcome 1, analysis 1]; Event rate = 12.3, 95% CI 2-sided [8.1 to 17.2] — Event and CI estimated using Kaplan-Meier method

25. Secondary Outcome: FDA Clearance Cohort: Rate of All Intracranial Hemorrhage (ICH)
Description: Independent core lab adjudicated rate of all ICH at 24-hour post-procedure
Time Frame: 24-hour post-procedure
Population: The FDA Clearance Cohort comprises participants in whom concomitant dual aspiration was used (e.g., 0.088" ID and a smaller ID catheter). One participant is missing imaging for core lab adjudication.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 210
Participants | 42

26. Secondary Outcome: FDA Clearance Cohort: Rate of Embolization in New Territory (ENT)
Description: as for outcome 15
Time Frame: End of procedure to 24-hour post-procedure
Population: The FDA Clearance Cohort comprises participants in whom concomitant dual aspiration was used (e.g., 0.088" ID and a smaller ID catheter). Participants with completed ENT forms are evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 200
Participants | 2

27. Secondary Outcome: FDA Clearance Cohort: Rate of Serious Adverse Device Effects (SADEs)
Description: Independent Safety Board adjudicated device-related serious adverse device events within 90 days post-procedure
Time Frame: 90-days post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 211
Participants | 3

28. Secondary Outcome: FDA Clearance Cohort: Rate of Serious Adverse Events
Description: All serious adverse events through 90 days post-procedure.
Time Frame: 90-days post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 211
Participants | 74

29. Secondary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Time to Achieve mTICI Score ≥ 2b
Description: The time from groin puncture to mTICI (modified treatment in cerebral infarction) score ≥ 2b flow.
  mTICI range: 0 to 3; higher score means better reperfusion
Time Frame: Intraprocedural
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 145
minutes | 18 [12 to 27.3]

30. Secondary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of mTICI Score 3 Reperfusion
Description: as for outcome 8
Time Frame: Intraprocedural
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 145
Participants | 46

31. Secondary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of First Pass Success
Description: Independent core lab-adjudicated modified treatment in cerebral infarction (mTICI) score ≥2b after the first pass with the study device
  mTICI range: 0 to 3; higher score means better reperfusion
Time Frame: Intraprocedural
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 145
Participants | 87

32. Secondary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of mTICI Score 2c Reperfusion
Description: as for outcome 21
Time Frame: Intraprocedural
Population: Post thrombectomy imaging available for core lab adjudication
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 145
Participants | 84

33. Secondary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of Functional Independence
Description: as for outcome 11
Time Frame: 90-days post-procedure
Population: Subjects with completed mRS assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 134
Participants | 67

34. Secondary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Quality of Life Assessment
Description: as for outcome 12
Time Frame: 90-days post-procedure
Population: FDA Clearance Cohort - Covariate Analysis for Distal ICA/M1 Occlusions in subjects completing SIS assesment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 96
score on a scale
  Overall Recovery | 69 (27)
  Strength | 69.4 (28.4)
  Memory and Thinking | 76.5 (23.8)
  Emotion | 78.6 (17.6)
  Communication | 84.7 (23.6)
  Activities of Daily Living or Instrumental Activities of Daily Living | 74.6 (29.8)
  Mobility | 70 (30)
  Hand Function | 66.4 (36.9)
  Participation/Role Function | 68.5 (30.9)

35. Secondary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of All-Cause Mortality
Description: Rate of 90-day all-cause mortality
Time Frame: 90-days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 146
Participants | 21

36. Secondary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of All Intracranial Hemorrhage (ICH)
Description: Independent core lab adjudicated rate of all ICH at 24-hour post-procedure
Time Frame: 24-hour post-procedure
Population: FDA Clearance Cohort - Covariate Analysis for Distal ICA/M1 Occlusions; Based on available imaging: Procedural imaging was not available for one (1) participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 145
Participants | 29

37. Secondary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of Embolization in New Territory (ENT)
Description: as for outcome 15
Time Frame: End of procedure to 24-hour post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 136
Participants | 2

38. Secondary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of Serious Adverse Device Effects (SADEs)
Description: Independent Safety Board adjudicated device-related serious adverse device events within 90 days post-procedure
Time Frame: 90-days post-procedure
Population: FDA Clearance Cohort - Covariate Analysis for Distal ICA/M1 Occlusions
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 146
Participants | 3

39. Secondary Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of Serious Adverse Events
Description: All serious adverse events through 90 days post-procedure
Time Frame: 90-days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 146
Participants | 54

40. Post Hoc Outcome: ITT Cohort: Rate of Rescue to Achieve mTICI Score ≥2b
Description: Use of additional devices to achieve core lab adjudicated mTICI score ≥2b
Time Frame: Intraprocedural
Population: Patients in whom mTICI score ≥2b was achieved
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 238
Participants | 13

41. Post Hoc Outcome: FDA Clearance Cohort: Rate of Rescue to Achieve mTICI Score ≥ 2b
Description: Use of additional devices to achieve mTICI Score ≥ 2b
Time Frame: Intraprocedural
Population: Participants in whom mTICI Score ≥ 2b was achieved
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 192
Participants | 9

42. Post Hoc Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of Rescue to Achieve mTICI Score ≥ 2b
Description: Use of additional devices to achieve mTICI Score ≥ 2b
  mTICI range: 0 to 3; higher score means better reperfusion
Time Frame: Intraprocedural
Population: Participants in whom mTICI Score ≥ 2b was achieved
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 135
Participants | 5

43. Post Hoc Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of mTICI Score ≥2b After All Study Device Passes
Description: Independent core lab-adjudicated reperfusion success, defined as modified treatment in cerebral infarction (mTICI) score ≥2b, after all passes with the study device. Additional device use after mTICI score ≥2b was achieved with study device was not imputed as failure.
Time Frame: Intraprocedural
Population: FDA Clearance Cohort - Covariate Analysis for Distal ICA/M1 Occlusions
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 145
Participants | 130

44. Post Hoc Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of mTICI Score ≥2b After All Study Device Passes, Additional Device Use Was Imputed as Failure
Description: Independent core lab-adjudicated reperfusion success, defined as modified treatment in cerebral infarction (mTICI) score ≥2b, after all passes with the study device. Additional device use after mTICI score ≥2b was achieved with study device was imputed as failure.
Time Frame: Intraprocedural
Population: FDA Clearance Cohort - Covariate Analysis for Distal ICA/M1 Occlusions
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 145
Participants | 126

45. Post Hoc Outcome: FDA Clearance Cohort for Distal ICA/M1 Occlusions: Rate of mTICI Score ≥2b at the End of the Procedure
Description: Independent core lab-adjudicated reperfusion success, defined as modified treatment in cerebral infarction (mTICI) score ≥2 at the end of the procedure, including rescue therapy with non-study devices
Time Frame: Intraprocedural
Population: FDA Clearance Cohort - Covariate Analysis for Distal ICA/M1 Occlusions
Measure: Count of Participants; unit: Participants
Arm/Group | Zoom Reperfusion System
Number analyzed (Participants) | 145
Participants | 135

ADVERSE EVENTS:
Time Frame: Throughout 90 days post-procedure
Arm/Group | Zoom Reperfusion System
All-Cause Mortality (participants affected / at risk) | 33/260
Serious Adverse Events (participants affected / at risk) | 95/260
Other Adverse Events (participants affected / at risk) | 165/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoom Reperfusion System (N=260)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Cardiac arrest (Cardiac disorders) | 4 (4)
Cardiac failure (Cardiac disorders) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4)
Pneumonia (Infections and infestations) | 7 (7)
Urinary tract infection (Infections and infestations) | 4 (4)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) — All groin pseudoaneurysms
Vessel perforation (Injury, poisoning and procedural complications) | 3 (3)
Brain oedema (Nervous system disorders) | 8 (8)
Cerebral artery occlusion (Nervous system disorders) | 3 (3)
Cerebral artery restenosis (Nervous system disorders) | 4 (4)
Cerebral haemorrhage (Nervous system disorders) | 4 (4)
Cerebrovascular accident (Nervous system disorders) | 7 (7)
Haemorrhagic transformation stroke (Nervous system disorders) | 5 (5)
Seizure (Nervous system disorders) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoom Reperfusion System (N=260)
Anaemia (Blood and lymphatic system disorders) | 7 (7)
Leukocytosis (Blood and lymphatic system disorders) | 13 (13)
Atrial fibrillation (Cardiac disorders) | 20 (20)
Dysphagia (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 8 (8)
Pneumonia (Infections and infestations) | 14 (14)
Urinary tract infection (Infections and infestations) | 16 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 7 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6)
Hypernatraemia (Metabolism and nutrition disorders) | 11 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (15)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (6)
Brain oedema (Nervous system disorders) | 6 (6)
Cerebral haemorrhage (Nervous system disorders) | 10 (10)
Cerebral microhaemorrhage (Nervous system disorders) | 6 (6)
Cerebral vasoconstriction (Nervous system disorders) | 7 (7)
Haemorrhage intracranial (Nervous system disorders) | 14 (14)
Haemorrhagic transformation stroke (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 10 (10)
Seizure (Nervous system disorders) | 6 (6)
Subarachnoid haemorrhage (Nervous system disorders) | 8 (8)
Agitation (Psychiatric disorders) | 8 (8)
Acute kidney injury (Renal and urinary disorders) | 13 (13)
Urinary retention (Renal and urinary disorders) | 15 (15)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Hypertension (Vascular disorders) | 11 (11)
Hypotension (Vascular disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT04129125/Prot_SAP_001.pdf